CLINICAL TRIAL: NCT02490605
Title: Effect of the Use of an Occlusal Plate on the Postural Alignment and Balance of Individuals With Signs and Symptoms of Temporomandibular Joint Disorder
Brief Title: Effect of the Use of an Occlusal Plate on the Postural Alignment
Acronym: Simone
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Maria Luiza Moreira Arantes Frigerio (Unknown)
Responsible Party: Principal Investigator, Simone Saldanha Ignacio de Oliveira, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Simone
Record Dates: First submitted 2015-06-05; First posted 2015-07-07 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Temporomandibular Joint Disorders
Keywords: Postural balance; Temporomandibular disorders; Splints
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- occlusal plate group (Experimental): The sample group will receive an occlusal plate with criteria for occlusal stability (simultaneous, bilateral contacts with an absence of interference in the canine and anterior guides). The occlusal plate will be made from "Vacuum Form" acetate with a thickness of 1.5 mm; the simultaneous, bilateral, occlusal contacts and the canine and anterior guides will be obtained by way of autopolymerizable, acrylic resin with the mandible in a centric relationship.
  Interventions: Procedure: occlusal plate group; Procedure: therapeutic exercises
- therapeutic exercises (Active Comparator): The control group will only receive orientation to do physiotherapeutic exercises seeking to correctly position the mandible in the resting position (maxillar teeth should be approximately 2 mm away from the mandibular teeth) while the tip of the tongue is positioned and accommodated on the roof of the mouth over the incisive papilla on the hard palate (without touching the teeth). The exercise will consist of repeatedly opening the mouth with the tongue cleaving to the roof of the mouth, 3 times per day, each period consisting of 3 sets with 15 repetitions.
  Interventions: Procedure: therapeutic exercises

INTERVENTIONS:
Procedure: occlusal plate group — occlusal plate with criteria for occlusal stability (simultaneous, bilateral contacts with an absence of interference in the canine and anterior guides
  Arms: occlusal plate group
Procedure: therapeutic exercises — The exercise will consist of the movement of repeatedly opening the mouth with the tongue cleaving to the "roof of the mouth" 3 times per day with each period consists of of 3 sets with 15 repetitions

SUMMARY:
The possible relationship between posture and instability of the masticatory muscles related to occlusion thus becomes the reason, the objective of this study. In this way, it will be possible to evaluate both postural alignment and postural balance in patients with signs and symptoms of temporomandibular joint disorder before and after the use of an occlusal plate. Our research will take place at the School of Odontology of the University of São Paulo in the clinics of the Occlusion and TMJ Services (SOA) and of the Envelhecer Sorrindo program, and the data will be collected in the Biophysics Laboratory of the School of Physical Education and Sports of the University of São Paulo. The population studies will be made up of 120 patients, 60 being part of the sample and the other 60 in the control group. All the patients in this study are over 20 years of age and are of both genders; the research criteria will be diagnosed by way of filling out the questionnaire of the RDC-TMD and complemented by way of diagnostic imaging via MRI of the temporomandibular joint. The study will be a clinical, randomized, controlled, prospective study and intervention. After the subjects' alignment is evaluated by way of photographs and their postural balance by way of a force platform, the group will the randomized; the sample group will receive an occlusal plate with criteria for occlusal stability (simultaneous, bilateral contacts with an absence of interference in the canine and anterior guides). The occlusal plate will be made from "Vacuum Form" acetate with a thickness of 1.5 mm; the simultaneous, bilateral, occlusal contacts and the canine and anterior guides will be obtained by way of autopolymerizable, acrylic resin with the mandible in a centric relationship. The occlusal plate will be controlled weekly. The control group will only receive orientation to do physiotherapeutic exercises seeking to correctly position the mandible in the resting position (maxillar teeth should be approximately 2 mm away from the mandibular teeth) while the tip of the tongue is positioned and accommodated on the roof of the mouth over the incisive papilla on the hard palate (without touching the teeth). The exercise will consist of repeatedly opening the mouth with the tongue cleaving to the roof of the mouth, 3 times per day, each period consisting of 3 sets with 15 repetitions. After 3 months, the two groups will be re-evaluated in terms of postural alignment and balance.

DETAILED DESCRIPTION:
The data will undergo the pertinent statistical treatment. The supposition is that those who undergo re-education of their neuromuscular system will see improvement in their coordination and understanding in relationship to TMJ, re-establishing the function by way of the occlusal stability.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are more than 20 years old,
* Both genders,
* Patients who present signs and symptoms of TMD identified by way of filling out the questionnaire of the RDC-TMD (Diagnostic Research Criteria) complemented by way of diagnostic imaging via an MRI of the temporomandibular joint.
* Patients who have their natural teeth, allowing for the use of partial, removable, Class-III Kennedy prostheses with small and medium spaces (up to 3 elements), having as a criteria posterior control (patients with partial, removable prostheses without presenting any type of compression marks or lesions under the structure, points of trauma indicated by redness of the mucosa, and verification of simultaneous, bilateral contacts) (Stegun; Costa, 2000).
* Patients who undergo the MRI of the temporomandibular joint at the time of the evaluation.

Exclusion Criteria:

* Patients entirely without unimaxillar and bimaxillar teeth,
* Patients with a dislocated disc without reduction,
* Patients with a history of cervical macrotraumas,
* Patients who continually use analgesics and anti-inflammatories, and/or medications that might effect their balance,
* Patients with compromised vision without corrections,
* Patients with neurological alterations,
* Patients with a history of falls,
* Patients with diabetes accompanied by sensitive neuropathies,
* Patients who complain of labyrinthitis.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2015-07; Primary Completion 2015-09 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
To investigate the effects of the use of occlusal splint over postural alignment | twelve weeks
  alignment will be evaluate by means 32 anatomic points to evaluate posture via the SAPO protocol, which is based on the evaluation of the subject in four photographic views (anterior front, posterior front, right side, and left side)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Luiza MA Frigerio, PhD, Principal Investigator — Universidade de São Paulo - Brazil - 05508-900
Locations (1):
- Universidade de São Paulo, São Paulo, São Paulo, Brazil